CLINICAL TRIAL: NCT03751384
Title: Fish Oil Supplementation in Cancer Patients - Capsules or in Nutritional Supplements. A Controlled Trial of Compliance.
Brief Title: Improvement of Compliance for High Doses of EPA Amongst Patients With Colorectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Jens Rikardt Andersen, Associated Professor, University of Copenhagen
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: H-15000693
Record Dates: First submitted 2018-11-16; First posted 2018-11-23 (Actual); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Compliance; Abdominal Cancer
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Intervention Model Description: Allocation, not randomized
Who Masked: Outcomes Assessor
Masking Description: pseudo-anonymized

ARMS (2):
- Capsules (Experimental): Dietary Supplement: Möllers Omega-3 Ekstra Sterk
  Interventions: Dietary Supplement: Möllers Omega-3 Ekstra Sterk
- Drink (Active Comparator): Dietary Supplement: Nutrifriend Cachexia
  Interventions: Dietary Supplement: Nutrifriend Cachexia

INTERVENTIONS:
Dietary Supplement: Möllers Omega-3 Ekstra Sterk
  Arms: Capsules
Dietary Supplement: Nutrifriend Cachexia
  Arms: Drink

SUMMARY:
Several studies indicate beneficial effects of eicosapentanoic acid (EPA) on cancer cachexia. However, compliance is generally low. This case control study is conducted in order to investigate if compliance depends upon the physical properties of the supplement (capsules vs. drinks). In order to further investigate how compliance can be improved, a possible correlation between sideeffects and rate of increased polyunsaturated fatty acid concentration in blood is also tested

DETAILED DESCRIPTION:
Patients with abdominal cancer in active chemotherapeutic were allocated to either EPA in an oral nutritional drink (commercial) or capsules with fish oil. The dose of EPA was the same in both groups, and diets were adjusted as iso-caloric. Compliance to the fish oil treatment was the primary outcome. Blood concentrations of EPA secondary.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving chemotherapy on Rigshospitalet due to colorectal cancer
* Not terminally ill
* Subjects must be18 years of age (or older)

Exclusion Criteria:

* Subjects who do not read/speak/understand Danish
* Familial hypercholesterolemia
* Predialytic patients (GFR < 15 ml/min/1,73 m2 or creatinine ≥ 500 mmol/L)
* Use of blood thinners
* Bleeder's disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2015-05-18 (Actual); Primary Completion 2017-09-25 (Actual); Study Completion 2018-11-10 (Actual)

PRIMARY OUTCOMES:
Compliance | 4 weeks
  Number of Capsules and bottles counted

SECONDARY OUTCOMES:
Erythrocyte concentration of EPA | 4 weeks
  Concentration measured on isolated erythrocytes

CONTACTS AND LOCATIONS:
Overall Officials: Jens R Andersen, Principal Investigator — University of Copenhagen
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schmidt N, Moller G, Baeksgaard L, Osterlind K, Stark KD, Lauritzen L, Andersen JR. Fish oil supplementation in cancer patients. Capsules or nutritional drink supplements? A controlled study of compliance. Clin Nutr ESPEN. 2020 Feb;35:63-68. doi: 10.1016/j.clnesp.2019.12.004. Epub 2020 Jan 3. PMID 31987122